CLINICAL TRIAL: NCT04527562
Title: Colchicine in Moderate Symptomatic COVID-19 Patients: Double Blind, Randomized, Placebo Controlled Trial to Observe the Efficacy
Brief Title: Colchicine in Moderate Symptomatic COVID-19 Patients
Acronym: COLCOVIDBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dhaka Medical College (Other)
Responsible Party: Principal Investigator, Dr. Md. Motlabur Rahman, Associate Professor, Department of Medicine, Dhaka Medical College
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: U1111-1255-3541
Record Dates: First submitted 2020-08-25; First posted 2020-08-26 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Covid19
Keywords: Covid 19; Colchicine
MeSH Terms: conditions — COVID-19 | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TRAETMENT GROUP (Active Comparator): Participants in the colchicine treatment group will be given a starting dose of 1.2 mg of Colchicine (2 tablets of 0.6 mg )single or 12 hourly divided dose. After that, they will take colchicine 0.6mg daily for 13 days. If they develop gastro intestinal side effects e.g abdominal pain, burning, vomiting, diarrhea, omeprazole and antiemetic will be prescribed.
  Interventions: Drug: Colchicine
- CONTROL /PLACEBO GROUP (Placebo Comparator): COVID-19 Patients in this arm will receive standard COVID-19 treatment according to national guidelines of Bangladesh and will receive placebo.
  Standard care of enrolled study patients will consist:
  1. Isolation facility
  2. Symptomatic treatment with Paracetamol, Fexofenadine
  3. Steam inhalation/Gurgle of Lukewarm water.
  4. Ensuring of hand wash (20 seconds each time) and ideally wearing mask.
  5. Monitoring by the attending nurses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine — Participants in this group will be given a starting dose of 1.2 mg of Colchicine (2 tablets of 0.6 mg )single or 12 hourly divided dose. After that, they will take colchicine 0.6mg daily for 13 days. If they develop gastro intestinal side effects e.g abdominal pain, burning, vomiting, diarrhea, omeprazole and antiemetic will be prescribed. Supportive care and treatment will also be given.
  Arms: TRAETMENT GROUP
Drug: Placebo — Participants in this group will be given a starting dose of 2 tablets of Placebo, single or 12 hourly divided dose. After that, they will take one placebo tablet daily for 13 days.Placebo tablet will be identical with the Colchicine tablet. If patients develop gastro intestinal side effects e.g abdominal pain, burning, vomiting, diarrhea, omeprazole and antiemetic will be prescribed. Supportive care and treatment will also be given.
  Arms: CONTROL /PLACEBO GROUP

SUMMARY:
This is a prospective, double blind, randomized, placebo controlled clinical trial. The participants will be randomized into two groups (group A and group B). Patients of group-A are the treatment group. They will be treated with optimal treatment based on the algorithm proposed in National Guidelines on Clinical Management of Coronavirus Disease 2019 (Covid-19) Version 7.0, 28 May 2020, along with Colchicine for 14 days. The patients in group-B will be controlled group. They will be treated with optimal treatment based on the algorithm proposed in National Guideline along with a placebo.

ELIGIBILITY:
Inclusion criteria:

* Males and females of least 18 years of age and can swallow tablets
* Competent and willing to provide informed consent
* Patient must have received a diagnosis of COVID-19 infection with positive RT-PCR for SARS CoV-2 within the last 3 days
* Patients with moderate symptoms (According to National Guidelines on Clinical Management of Coronavirus Disease 2019 (COVID- 19).Version 7.0 .2020, DGHS, MOHFW, Government of the People's Republic of Bangladesh). Following features of moderate covid-19 must be present-

  1. Fever or history of fever
  2. Cough and /or Shortness of breath
  3. Oxygen saturation 94% or more
  4. Pneumonia -pulmonary consolidations on chest imaging (chest x ray or CT scan of chest) involving less than 50%of lungs
  5. CRB 65 score 0

Exclusion criteria:

* Pregnancy and breast-feeding
* Known hypersensitivity to colchicine
* Known chronic illness e.g hepatic failure, chronic kidney disease (eGFR<30ml/min), decompensated heart failure, long QT syndrome (QTc >450 msec.)
* Patient with inflammatory bowel disease (Crohn's disease or ulcerative colitis), chronic diarrhea or malabsorption
* Patient currently taking colchicine for other indications (mainly chronic indications represented by Familial Mediterranean Fever or gout)
* Patient undergoing chemotherapy for cancer
* Patient is considered by the investigator, for any reason, to be an unsuitable candidate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Time to develop clinical deterioration, defined as the time from randomization to a deterioration of two points (from the status at randomization) on a Seven-category ordinal scale. | 14 days following randomization
  Seven-category ordinal scale. The scale is recommended by the WHO R&D Blueprint expert group. The seven-category ordinal scale consisted of the following categories: 1, not hospitalized with resumption of normal activities; 2, not hospitalized, but unable to resume normal activities; 3, hospitalized, not requiring supplemental oxygen; 4, hospitalized, requiring supplemental oxygen; 5, hospitalized, requiring nasal high-flow oxygen therapy, noninvasive mechanical ventilation, or both; 6, hospitalized, requiring ECMO, invasive mechanical ventilation, or both; and 7, death

SECONDARY OUTCOMES:
Length of hospital stay | 14 days following randomization
  Days from date of enrollment to date of discharge
Number of participant requiring increased amount of supplemental oxygen | 14 days following randomization
  Proportion of participants who required oxygen supplementation
Number of participants requiring mechanical ventilation | 14 days following randomization
  Proportion of participants who required mechanical ventilation
Number of participants who die | 14 days following randomization
  Proportion of participants who die from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Mujibur Rahman, MBBS,MD,FCPS, Study Chair — Professor and Head, Department of Medicine; Motlabur Rahman, MBBS, FCPS,FACP, Principal Investigator — Associate Professor, Department of Medicine
Locations (1):
- Dhaka Medical College Hospital, Dhaka-1000, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rahman M, Datta PK, Islam K, Haque M, Mahmud R, Mallik U, Hasan P, Haque M, Faruq I, Sharif M, Ratul RH, Azad KAK, Miah T, Rahman MM. Efficacy of colchicine in patients with moderate COVID-19: A double-blinded, randomized, placebo-controlled trial. PLoS One. 2022 Nov 16;17(11):e0277790. doi: 10.1371/journal.pone.0277790. eCollection 2022. PMID 36383611